CLINICAL TRIAL: NCT05615441
Title: Effect of Nociception Level Monitoring During Remimazolam-based Total Intravenous Anesthesia on Intraoperative Opioid Requirements and Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2022-1155
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Adult Patients Aged 19-64, Scheduled for Elective Arthroscopic Knee Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI-guided (Active Comparator): Patients receiving remimazolam-based total intravenous general anesthesia with nociception monitoring with the ANI monitor
  Interventions: Device: Analgesia Nociception Index monitor
- Standard (Experimental): Patients receiving remimazolam-based total intravenous general anesthesia based on hemodynamic variables and without ANI nociception monitoring
  Interventions: Device: Standard monitoring

INTERVENTIONS:
Device: Analgesia Nociception Index monitor — Patients will receive remimazolam-based total intravenous general anesthesia with nociception monitoring with the ANI monitor
  Arms: ANI-guided
Device: Standard monitoring — Patients will receive remimazolam-based total intravenous general anesthesia based on hemodynamic monitoring and without nociception monitoring
  Arms: Standard

SUMMARY:
This study aims to investigate whether the use of nociception monitoring during general anesthesia with remimazolam-based total intravenous anesthesia has an effect on intraoperative opioid requirements and postoperative pain. This study is a randomized trial with a 50% probability of being assigned to either group. Randomization will be done by an anesthesiologist not involved in anesthesia or postoperative outcome assessment. Patients and the investigator in charge of postoperative outcomes assessment will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

Adult patients between 19 and 64 years of age, ASA class I~III, scheduled for arthroscopic knee surgeryunder general anesthesia.

Exclusion Criteria:

Patient refusal, patients unable to read consent form, active URI or uncontrolled asthma, pneumonia, history of allergies to benzodiazepines, decreased liver or kidney function, heart failure of ejection fraction<55%, pregnant or breastfeeding patients, history of substance abuse/addiction

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil requirement | Within the intraoperative period
  Intraoperative remifentanil requirements will be collected as primary outcome as µg/kg/min

CONTACTS AND LOCATIONS:
Overall Officials: Seokyung Shin, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No